CLINICAL TRIAL: NCT06339866
Title: Effect of Two Different Video Showings on Pain and Anxiety in Children Undergoing Adenotonsillectomy: A Randomized Controlled Study
Brief Title: The Effect of Two Different Video Showings on Pain and Anxiety in Children Undergoing Adenotonsillectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, mihriye koca, Master student, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: E16734702
Record Dates: First submitted 2023-10-04; First posted 2024-04-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pain After Adenotonsillectomy
Keywords: pain,adenotonsillectomy,anxiety,children

STUDY DESIGN:
Intervention Model Description: The population of the research will be all patients who had adenotonsillectomy surgery between the ages of 6-12 in the Ear Nose and Throat Service of Zonguldak Bülent Ecevit University Hospital, and the sample will be all patients who had adenotonsillectomy surgery between the specified dates and who meet the inclusion criteria.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The control group will follow the routine plan of the ward without any intervention planned.
- Educational animation group (Experimental): After the patients in this group arrive at the ward (after adenotonsillectomy), the Wong Baker pain scale and Child Anxiety Scale-Status (CAS-D) will be filled out by three observers (clinic nurse, parent and child) before the educational animated movie (before analgesic application) containing the surgical process at the 3rd hour (after adenotonsillectomy) and the animation will be watched behind it, and at the end, the same scales will be filled out again by three observers and the patient's pain and anxiety level will be evaluated.
  Interventions: Other: The Effect of Two Different Video Interventions on Pain and Anxiety in Children with Adenotonsillectomy: A Randomized Controlled Study
- Cartoon series group (Experimental): In this group, the Wong Baker pain scale and Child Anxiety Scale-Disposition (CAS-D) will be filled out by three observers before watching cartoons at the 3rd hour post op (before analgesic administration), and the scales will be filled out again after the cartoon and anxiety and pain levels will be evaluated.
  Interventions: Other: The Effect of Two Different Video Interventions on Pain and Anxiety in Children with Adenotonsillectomy: A Randomized Controlled Study

INTERVENTIONS:
Other: The Effect of Two Different Video Interventions on Pain and Anxiety in Children with Adenotonsillectomy: A Randomized Controlled Study — The population of the study will be all patients who had adenotonsillectomy surgery between the ages of 6-12 in the Ear Nose and Throat Service of Zonguldak Bülent Ecevit University Hospital, and the sample will be all patients who had adenotonsillectomy surgery between the specified dates and who meet the inclusion criteria.
  Arms: Cartoon series group; Educational animation group

SUMMARY:
Purpose of the Research: The purpose of the research is to examine the effect of two different video presentations on pain and anxiety in children undergoing adenotonsillectomy.

Type of Research It is planned as a randomized controlled interventional type study to examine the effects of two different video presentations on pain and anxiety in children undergoing adenotonsillectomy.

DETAILED DESCRIPTION:
Technology is an indispensable part of our age and daily life . When we look at the research, it is seen that educational interventional preparation programs increase the harmony between both children, parents and health professionals. The increase in children's self-control and the elimination of unrealistic expectations may be related to the trust in healthcare professionals. Studies indicate that educational video animations are the most effective non-pharmacological method in reducing anxiety . Video animations will be useful for children because they create sound and images. It is believed that video animations with educational content that are understandable to children are essential for children's education. It is believed that animation shown to children will reduce their anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 6-12
* Having adenotonsillectomy surgery
* Signing the informed consent form by the patient's legal guardian

Exclusion Criteria:

* Not being between the ages of 6-12
* Not having adenotonsillectomy surgery
* Failure to sign the enformel consent form by the patient's legal guardian

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
After the intervention, the mean score of the children in the postoperative animation and cartoon group on the Wong Baker Pain Rating Scale will be lower than those in the control group. | 6 months
  The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst." As the score increases, the child's pain improves.

SECONDARY OUTCOMES:
After the intervention, the mean score of the Children's Anxiety Scale-Stability score of the children in the postoperative animation and cartoon group will be less than those in the control group. | 6 months
  The CASS is configured as a thermometer, including a bulb chamber at the bottom and horizontal lines upwards. Each horizontal line represents one score and the thermometer has 10 points. The bulb chamber at the bottom has 0 points and indicates no anxiety. As horizontal lines rise upwards, it is interpreted as an increase in anxiety. The highest score is 10, referring to the highest anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Mihriye, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: THE EFFECT OF A CARTOON AND AN INFORMATION VIDEO ABOUT INTRAVENOUS INSERTION ON PAIN AND FEAR IN CHILDREN AGED 6 TO 12 YEARS IN THE PEDIATRIC EMERGENCY UNIT: A RANDOMIZED CONTROLLED TRIAL — https://pubmed.ncbi.nlm.nih.gov/32690314/